CLINICAL TRIAL: NCT03862196
Title: Efficacy of an Intervention With Text Messaging to Improve Early Retention in HIV Care for People With HIV Who Receive Treatment at VIA LIBRE
Brief Title: Efficacy of SMS to Improve Early Retention in HIV Care for PLWH in Lima
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NGO Via Libre (Other)
Responsible Party: Principal Investigator, ROBINSON CABELLO, Executive Director, NGO Via Libre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NGOViaLibre
Record Dates: First submitted 2018-11-28; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: prevention; retention; mHealth

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot study with a parallel 2-arm design.The intervention arm will receive 2 tailored text messages weekly from a trained counselor during 3 months. The control arm will receive the standard of care, which consists of pre and post counseling after the HIV diagnosis and referral to a health facility to start antiretroviral treatment.
Who Masked: Care Provider
Masking Description: After consenting, participants will be randomly assigned to the intervention or control with a 1:1 ratio and random block sizes of 2 and 4 using computer generated random numbers. Block sizes will not be disclosed. Allocations will be sealed in individual, sequentially numbered opaque envelopes. The RECRUITER, who will be masked to the group assignment, will give instructions to all participants on how they should interact if they start receiving SMS. After completing the baseline survey, one of the principal investigators will assign the participant to a group by opening the corresponding envelope. The PI will report to one of trained providers in charge of delivering the intervention (different from recruiters) when a new participant of the intervention arm is enrolled. Because of the nature of the participation, providers and participants will not be masked to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive 2 tailored text messages weekly from a trained counselor during 3 months.
  Interventions: Behavioral: Tailored text messages to improve retention in HIV care
- Control (No Intervention): Participants will receive standard of care: pre and post counseling after being diagnosed with HIV

INTERVENTIONS:
Behavioral: Tailored text messages to improve retention in HIV care — Trained counselors will deliver the text messages. After a block randomization, the trained counselor (a nurse) will send the first welcoming message to participants in the intervention arm. The nurse will send 2 tailored text messages per week. In addition 2 to 4 days before an appointment, the nurse will send a message reminder. In addition, the nurse will have bilateral communication with participants using text messages according to their needs. The participants of the intervention arm will interact with the nurse during 3 months with a semi-structured strategy, that is, with template text messages (predesigned) and open messages (for which the nurse will be trained). Three and six months after started the intervention the variables of interest will be assessed.
  Arms: Intervention

SUMMARY:
Randomized controlled study that will evaluate the effect of a text message-based strategy to improve retention in HIV care.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study with a parallel 2-arm design. It will evaluate the effect of a text message-based strategy to improve retention in HIV care at the study clinic, compared to the standard of care. Trained counselors will deliver the text messages. After a block randomization, the trained counselor (a nurse) will send the first welcoming message to participants in the intervention arm. The nurse will send 2 tailored text messages per week. In addition 2 to 4 days before an appointment, the nurse will send a message reminder. In addition, the nurse will have bilateral communication with participants using text messages according to their needs. The participants of the intervention arm will interact with the nurse during 3 months with a semi-structured strategy, that is, with template text messages (predesigned) and open messages (for which the nurse will be trained). Three and six months after started the intervention the variables of interest will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years old or older.
* Linked to HIV care at the study clinic.
* Have a cell phone.
* Diagnosed at the study clinic of referred from other center to start ART.
* Give consent to participate.

Exclusion Criteria:

* Enrolled in other HIV study using text messages.
* Have started ART.
* Enrolled in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-04-11 (Estimated); Study Completion 2019-08-07 (Estimated)

PRIMARY OUTCOMES:
Retention in timely monitoring of viral load (VL) | 6 months
  Rate of participants with a second lab result of VL available 6 months after initiation of ART, verified using lab records

OTHER OUTCOMES:
Retention in HIV care | 3 months
  Rate of participants who attended the 2nd and 3rd appointments for HIV care at the study clinic, verified using medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Via Libre, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menacho L, Garcia PJ, Blas MM, Diaz G, Zunt JR. What Men Who Have Sex With Men in Peru Want in Internet-Based Sexual Health Information. J Homosex. 2018;65(7):934-946. doi: 10.1080/00918369.2017.1364939. Epub 2017 Sep 22. PMID 28820663
- [Background] AIDS by the numbers. UNAIDS, 2016. Retrieved from: http://www.unaids.org/sites/default/files/media_asset/AIDS-by-the-numbers2016_en.pdf
- [Background] UNAIDS country Peru report, 2016. Retrieved from: http://www.unaids.org/en/regionscountries/countries/peru
- [Background] Chow JY, Konda KA, Borquez A, Caballero P, Silva-Santisteban A, Klausner JD, Caceres CF. Peru's HIV care continuum among men who have sex with men and transgender women: opportunities to optimize treatment and prevention. Int J STD AIDS. 2016 Oct;27(12):1039-1048. doi: 10.1177/0956462416645727. Epub 2016 Apr 20. PMID 27099168
- [Background] Wolff MJ, Cortes CP, Mejia FA, Padgett D, Belaunzaran-Zamudio P, Grinsztejn B, Giganti MJ, McGowan CC, Rebeiro PF; Caribbean, Central and South America network for HIV epidemiology (CCASAnet). Evaluating the care cascade after antiretroviral therapy initiation in Latin America. Int J STD AIDS. 2018 Jan;29(1):4-12. doi: 10.1177/0956462417714094. Epub 2017 Jun 15. PMID 28618980
- [Background] Prevention gap report. UNAIDS, 2016. Retrieved from: http://www.unaids.org/sites/default/files/media_asset/2016-prevention-gapreport_en.pdf
- [Background] Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection: Recommendations for a Public Health Approach. 2nd edition. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK374294/ PMID 27466667
- [Background] Muessig KE, LeGrand S, Horvath KJ, Bauermeister JA, Hightow-Weidman LB. Recent mobile health interventions to support medication adherence among HIV-positive MSM. Curr Opin HIV AIDS. 2017 Sep;12(5):432-441. doi: 10.1097/COH.0000000000000401. PMID 28639990
- [Background] Rana AI, van den Berg JJ, Lamy E, Beckwith CG. Using a Mobile Health Intervention to Support HIV Treatment Adherence and Retention Among Patients at Risk for Disengaging with Care. AIDS Patient Care STDS. 2016 Apr;30(4):178-84. doi: 10.1089/apc.2016.0025. PMID 27028183
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Bayona E, Menacho L, Segura ER, Mburu G, Roman F, Tristan C, Bromley E, Cabello R. The Experiences of Newly Diagnosed Men Who Have Sex with Men Entering the HIV Care Cascade in Lima, Peru, 2015-2016: A Qualitative Analysis of Counselor-Participant Text Message Exchanges. Cyberpsychol Behav Soc Netw. 2017 Jun;20(6):389-396. doi: 10.1089/cyber.2016.0435. PMID 28622034
- [Background] Yu Y, Luo D, Chen X, Huang Z, Wang M, Xiao S. Medication adherence to antiretroviral therapy among newly treated people living with HIV. BMC Public Health. 2018 Jul 4;18(1):825. doi: 10.1186/s12889-018-5731-z. PMID 29973167
- [Background] Mannheimer S, Friedland G, Matts J, Child C, Chesney M. The consistency of adherence to antiretroviral therapy predicts biologic outcomes for human immunodeficiency virus-infected persons in clinical trials. Clin Infect Dis. 2002 Apr 15;34(8):1115-21. doi: 10.1086/339074. Epub 2002 Mar 11. PMID 11915001
- [Background] Menacho LA, Blas MM, Alva IE, Roberto Orellana E. Short Text Messages to Motivate HIV Testing Among Men Who have Sex with Men: A Qualitative Study in Lima, Peru. Open AIDS J. 2013 Apr 5;7:1-6. doi: 10.2174/1874613601307010001. Print 2013. PMID 23802032
- [Background] Young SD, Cumberland WG, Nianogo R, Menacho LA, Galea JT, Coates T. The HOPE social media intervention for global HIV prevention in Peru: a cluster randomised controlled trial. Lancet HIV. 2015 Jan;2(1):e27-32. doi: 10.1016/S2352-3018(14)00006-X. PMID 26236767

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT03862196/Prot_SAP_000.pdf